CLINICAL TRIAL: NCT05008328
Title: Feasibility of Live, Receptive Music Therapy for Patients Undergoing Spontaneous Breathing Trials: a Pilot Study
Brief Title: Feasibility of Music Therapy for Spontaneous Breathing Trials
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study team decided to conclude the study and report it as a feasibility study.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00110030
Record Dates: First submitted 2021-07-28; First posted 2021-08-17 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Spontaneous Breathing Trial; Intubation; Mechanical Ventilation; Music Therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Therapy plus Standard Care (Experimental): Music therapy intervention in addition to standard hospital care during an SBT.
  Interventions: Other: Music therapy plus standard care during an SBT
- Standard Care (Active Comparator): Standard hospital care during an SBT.
  Interventions: Procedure: Standard care during an SBT

INTERVENTIONS:
Other: Music therapy plus standard care during an SBT — If the participant is randomly assigned to standard care plus music therapy, a music therapist will enter the room five minutes prior to the start of the breathing trial and begin to play quiet music on a guitar. The nurse will reduce medicine to bring the participant to an alert state. The music therapist will introduce themselves and the music intervention, and will continue to play quiet guitar music and sing softly while the respiratory therapist begins the breathing trial. The music therapist will continue playing and singing for 20 minutes into the breathing trial.
  Arms: Music Therapy plus Standard Care
Procedure: Standard care during an SBT — The patient's nurse will reduce sedatives so the patient is alert and awake. The respiratory therapist will introduce themselves to the patient and inform them of the SBT, stating they will turn off the ventilator machine and allow the patient to breathe independently. The respiratory therapist will switch off the ventilator and leave the room. The respiratory therapist and nurse will both be available throughout the SBT, and the ventilator will automatically turn on if the patient stops breathing. The SBT will last for 30-60 minutes.
  Arms: Standard Care

SUMMARY:
In this study, the investigators will study music therapy for patients during breathing trials, a procedure performed in intensive care units. Participants will be assigned either to standard medical care or standard medical care plus music therapy. Participants have a 50/50 chance (like flipping a coin) of being in either group. In the music therapy group, a board-certified music therapist will sing softly with guitar accompaniment to provide music during the breathing trial. The music is in addition to the usual treatment provided by hospital staff. Participants in the standard medical care group will receive the usual medical care given by hospital staff members. Information will be collected from participant's charts and by observation of vital signs during the breathing trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18+
* Admitted to MUSC's Main Hospital medical intensive care unit (MICU) or Ashley River Tower medical-surgical intensive care unit (MSICU)
* Intubated and will undergo a spontaneous breathing trial

Exclusion Criteria:

* Patients who have had any prior SBTs
* Patients known to have a neurological injury
* Patients who are known to be deaf
* Patients whom (or whose LAR) are unable or unwilling to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of successful initial spontaneous breathing trials (SBTs) vs failed initial SBTs | Up to 48 hours after the participant's initial SBT.
  A successful SBT is defined as when a patient sustains at least 30 minutes without mechanical ventilator support, as deemed by the respiratory therapist in the participant's chart.
  A failed SBT is defined as when a patient requires mechanical ventilator support within 30 minutes of the start of the SBT, as deemed by the respiratory therapist.

SECONDARY OUTCOMES:
Mean minutes sustained off ventilator support for failed SBTs | Up to 48 hours after the participant's initial SBT.
  Total minutes sustained off ventilator support, as noted by respiratory therapist in the participant's chart.
Mean score of heart rate at points throughout SBT | At minute 0 of the SBT, 10 minutes into the SBT, and 30 minutes into the SBT
  Recording of patient's heart rate via observation of monitor at three points throughout the SBT
Mean score of respiratory rate at points throughout SBT | At minute 0 of the SBT, 10 minutes into the SBT, and 30 minutes into the SBT
  Recording of patient's respiratory rate via observation of monitor at three points throughout the SBT
Mean score of blood pressure at points throughout SBT | At minute 0 of the SBT, 10 minutes into the SBT, and 30 minutes into the SBT
  Recording of patient's blood pressure via observation of monitor at three points throughout the SBT
Mean score of agitation as assessed by the Richmond Agitation-Sedation Scale at points throughout SBT | At minute 0 of the SBT, 10 minutes into the SBT, and 30 minutes into the SBT
  * 4 Combative- Overtly combative, violent, immediate danger to staff
  * 3 Very agitated- Pulls or removes tube(s) or catheter(s); aggressive
  * 2 Agitated- Frequent non-purposeful movement, fights ventilator
  * 1 Restless- Anxious but movements not aggressive vigorous 0 Alert and calm
    * 1 Drowsy- Not fully alert, but has sustained awakening (eye opening/contact) to voice (>10 seconds)
    * 2 Light sedation- Briefly awakens with eye contact to voice (<10 seconds)
    * 3 Moderate sedation- Movement or eye opening to voice (but no eye contact)
    * 4 Deep sedation- No response to voice, but movement or eye opening to physical stimulation
    * 5 Unarousable- No response to voice or physical stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Macel Reising, MT-BC, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) may be shared with researchers at Appalachian State University where data analysis will occur, as the PI is currently a graduate student at that institution. Only de-identified data will go to App State; no protected health information (PHI) will leave Medical University of South Carolina (MUSC). De-identified data may be published as a master's thesis or in academic journals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data sharing will become available during October 2021 and will occur until May 2022.
Access Criteria: IPD will be shared with the PI's academic advisor for analysis of results with the purpose of writing a master's thesis paper.